CLINICAL TRIAL: NCT03584334
Title: Cohort Study Evaluating 18FDG PET for Early Identification of Tumor Exhaust for Immunotherapy in Patients With Locally Advanced or Metastatic Non-Small Cell Bronchopulmonary Carcinoma or Melanoma
Brief Title: 18FDG PET for Early Identification of Tumor Exhaust for Immunotherapy in Patients With Locally Advanced or Metastatic Non-Small Cell Bronchopulmonary Carcinoma or Melanoma
Acronym: FDG-IMMUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/77; 2018-A00915-50 (Other: ANSM ID RCB)
Record Dates: First submitted 2018-06-04; First posted 2018-07-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Bronchopulmonary Carcinoma or Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized, multi-center, diagnostic performance study of 18FDG PET for identification of early tumor escape to immunotherapy in patients with unresectable melanoma or Broncho-Pulmonary Carcinoma No to Advanced or Metastatic Small Cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18FDG PET (Other): Diagnostic performance of 18FDG PET for identification of early tumor escape to immunotherapy in patients with unresectable melanoma or Broncho-Pulmonary Carcinoma No to Advanced or Metastatic Small Cells
  Interventions: Radiation: 18FDG PET

INTERVENTIONS:
Radiation: 18FDG PET — Diagnostic performance of 18FDG PET for identification of early tumor escape to immunotherapy in patients with unresectable melanoma or Broncho-Pulmonary Carcinoma No to Advanced or Metastatic Small Cells

SUMMARY:
The hypothesis of this diagnostic performance study is that, for patients treated for immunotherapy-treated melanoma or NSCLC, some metabolic parameters of the 18FDG dual-point PET scan distinguish inflammatory pseudo-progression from tumor progression true and thus improve the evaluation of tumor response to immunotherapy

DETAILED DESCRIPTION:
The originality of this study is based on the stakes of the early prediction of resistance to immunotherapy (early therapeutic escapes, side effects, cost of treatment etc.).

No prospective study has been published to date on the value of 18FDG PET to distinguish between true tumor progression and pseudo-progression. Studies are therefore needed to define new criteria for evaluating the metabolic response specific to immunotherapy, as well as the optimal timing of the interim examination.

The goal is to conduct a transversal, non-randomized, prospective, multi-center, diagnostic performance study, harmonizing the moments of the 18FDG PET scans, acquisition conditions and interpretation criteria. The use of a dual-point acquisition in PET will also make it possible to judge the kinetics of 18FDG lesion capture (calculation of the 18FDG retention index on the late image) with the objective of highlighting PET criteria to distinguish between inflammatory pseudo-progression and true tumor progression in patients with unresectable melanoma or advanced or metastatic NSCLC. Other metabolic parameters will be studied, such as changes in tumor metabolic volume and binding intensities.

Finally, this study will include patients to assess the correlation between the metabolic tumor response observed after 7 weeks of immunotherapy, the morphological response after 3 months of treatment (RECIST v1.1 and i-RECIST) and survival overall at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years,
* Patients with unresectable melanoma or histologically proven, metastatic or locally advanced NSCLC,
* Indication of an immunotherapy treatment with nivolumab or pembrolizumab validated in multidisciplinary consultation team and prescribed as part of their marketing authorization, in first or second line of treatment,
* Performance Status 0 to 2,
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required,
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year,
* Male subjects should agree to use an adequate method of contraception or abstain from heterosexual activity starting with the first dose of study therapy through 6 months after the last dose of study therapy,
* Patient willing and able to provide written informed consent/assent for the trial,
* Patient affiliated with a health insurance system.

Exclusion Criteria:

* Age < 18 years,
* Contraindication to performing 18FDG PET scans: severe claustrophobia, unbalanced diabetes during PET examinations (fasting capillary blood glucose ≥ 11 mmol),
* Any participation in other biomedical studies related to the drug, medical devices or imaging techniques is prohibited except biomedical studies called overstudies (In case of doubt or questions about the patient's participation in a other clinical study, please contact the sponsor),
* Contraindication to nivolumab or pembrolizumab treatment,
* Patient with metastatic disease,
* History of thoracic irradiation or near / in the thoracic irradiation field,
* Patient who refuses to participate in the study or unable to agree,
* Patient currently receiving one or more treatments described in section 6.9 of the protocol,
* Contraindication to nivolumab or pembrolizumab treatment,
* People particularly vulnerable as defined in Articles L.1121-5 to -8 of the French Healthcare Code, including: person deprived of freedom by an administrative or judicial decision, adult being the object of a legal protection measure or outside a state to express their consent, pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Threshold of the 18FDG retention index (dual-point acquisition), from the first metabolic progression observed in 18FDG PET, to distinguish a true tumor progression from a pseudo-progression of inflammatory origin (leukocyte infiltrate) | 12 months
  ROC curve of the FDG retention index, defined on the dual-point PET acquisition, will be analysed to distinguish lesions in true progressions and lesions in inflammatory pseudo-progressions.

SECONDARY OUTCOMES:
PET criteria other than the 18FDG retention index to distinguish pseudo-progressions from true tumor progressions for new lesions: intensity of fixation (SUVpeak) and location of new lesions | 12 months
  It will be measured with absolute SUVpeak of new hyperfixing lesions
PET criteria other than the 18FDG retention index to distinguish pseudo-progressions from true tumor progressions for new lesions: intensity of fixation (SUVpeak) and location of new lesions | 12 months
  It will be measured with Percent change in fixation intensity of pre-existing lesions
PET criteria other than the 18FDG retention index to distinguish pseudo-progressions from true tumor progressions for new lesions: intensity of fixation (SUVpeak) and location of new lesions | 12 months
  It will be measured with Percentage of change in lesional tumor volume
PET criteria other than the 18FDG retention index to distinguish pseudo-progressions from true tumor progressions for new lesions: intensity of fixation (SUVpeak) and location of new lesions | 12 months
  It will be measured with Percentage of change in total Total Lesion
The incidence of inflammatory pseudo-progression compared to true tumor progressions, taking into account the impact of the primary tumor | 12 months
  Evaluation of the ratio between the lesions with an inflammatory pseudo-progression and those with a true tumor progression will be measured. A lesion and patient analysis will be performed
The incidence of inflammatory or infectious lesions diagnosed by 18FDG PET and their impact on clinical management | 12 months
  Frequency of inflammatory or infectious lesions accidentally diagnosed by PET will be measured
The incidence of inflammatory or infectious lesions diagnosed by 18FDG PET and their impact on clinical management | 12 months
  The number of these inflammatory diagnoses leading to specific management will be measured
The predictive value of the early metabolic response at 7 weeks on the morphological | 3 months
  Measurement of the association will be assessed with the early metabolic response at 7 weeks . The metabolic response will be evaluated according to PERCIST criteria.
The predictive value of the early metabolic response on metabolic responses at 3 months | 3 months
  Measurement of the association will be assessed with the morphological response at 3 months. The morphological response will be evaluated according to RECIST criteria v1.1 and i-RECIST in patients who have received the injection of iodine contrast product in PET scan
The prognostic value of the 7-week PET metabolic response on 12-month overall survival | 12 months
  To determine the delay between the date of inclusion and the date of death, overall survival will be measured at 12 months according to the changes in tumor metabolism on the interim PET at 7 weeks.
The prognostic value of the 3-month PET metabolic response on 12-month overall survival | 12 months
  To determine the delay between the date of inclusion and the date of death, overall survival will be measured at 12 months according to the changes in tumor metabolism on the interim PET at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- [Derived] Tricarico P, Chardin D, Martin N, Contu S, Hugonnet F, Otto J, Humbert O. Total metabolic tumor volume on 18F-FDG PET/CT is a game-changer for patients with metastatic lung cancer treated with immunotherapy. J Immunother Cancer. 2024 Apr 22;12(4):e007628. doi: 10.1136/jitc-2023-007628. PMID 38649279